CLINICAL TRIAL: NCT03671122
Title: PREFERS PREFERS (Preserved and Reduced Ejection Fraction Epidemiological Regional Study) Stockholm Heart Failure Study
Brief Title: PREFERS (Preserved and Reduced Ejection Fraction Epidemiological Regional Study) Stockholm Heart Failure Study
Acronym: PREFERS
Status: Completed | Type: Observational
Sponsor: Karolinska Institutet (Other)
Collaborators: The Swedish Research Council (Other Government); Region Stockholm (Other Government)
Responsible Party: Principal Investigator, Cecilia Linde, MD PhD Senior Professor, Karolinska Institutet
Other Study IDs: AZ, Molndal, Sweden grant 1377
Record Dates: First submitted 2018-09-09; First posted 2018-09-14 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Heart Failure, Diastolic; Heart Failure，Congestive
MeSH Terms: conditions — Heart Failure, Diastolic; Heart Failure | interventions — Echocardiography, Doppler; Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — In 500 of the included 1000 patients (CABG-PREFERS) needle biopsies are taken from the cardiac lateral wall of both the right and left ventricle before initiation of cardiac arrest and stored in -70 ∘C for histological and genetic analysis. Moreover biopsies are taken from the right atrial appendage (ample material), the right and left ventricular myocardium, as wellas from the internal mammary artery.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PREFERS main study: 500 patients with new onset heart failure will be characterized into those with HFpEFand HFrEF at baseline and undergo Cardiac imaging by Doppler echocardiography and cMRI, blood tests for biomarker analysis
  Interventions: Diagnostic Test: Cardiac imaging in the PREFERS and CABG PREFERS cohorts; Other: Biomarker analysis in the PREFERS and CABG PREFERS chorts
- CABG PREFERS: 500 Patients undergoing elective by pass surgery with or without diastolic or systolic dysfunction as Proxy for HFpEF and HFrEF will undergo Cardiac imaging by Doppler echocardiography and cMRI, blood tests for biomarker analysis and cardiac biopsies
  Interventions: Diagnostic Test: Cardiac imaging in the PREFERS and CABG PREFERS cohorts; Other: Biomarker analysis in the PREFERS and CABG PREFERS chorts; Procedure: Cardiac biopsies in the CABG PREFERS cohort

INTERVENTIONS:
Diagnostic Test: Cardiac imaging in the PREFERS and CABG PREFERS cohorts — performed at baseline and after 1 year
  Other Names: Doppler echocardiography and cMRI
Other: Biomarker analysis in the PREFERS and CABG PREFERS chorts — blood samples will be taken for biomarker analysis at baseline and after 1 year
  Other Names: blood samples
Procedure: Cardiac biopsies in the CABG PREFERS cohort — myocardial biopsies from the right trium the left and right ventricles will be taken during elective CABG
  Groups: CABG PREFERS

SUMMARY:
Heart failure (HF) with preserved (HFpEF) or reduced (HFrEF) ejection fraction is associated with poor prognosis and quality of life. While the incidence of HFrEF is declining and HF treatment is effective, HFpEF is increasing, with no established therapy. PREFERS Stockholm is an epidemiological study with the aim of improving clinical care and research in HF and to find new targets for drug treatment in HFpEF starting with a cardiac biopsy study in elective CABG patiens.

DETAILED DESCRIPTION:
Patients with new-onset HF (n = 2000) will be characterized at baseline and after 1-year follow-up by standardized protocols for clinical evaluation, echocardiography, and ECG. In one subset undergoing elective coronary bypass surgery (n = 100) and classified according to LV function, myocardial biopsies will be collected during surgery, and cardiac magnetic resonance (CMR) imaging will be performed at baseline and after 1 year. Blood and tissue samples will be stored in a biobank.We will characterize and compare new-onset HFpEF and HFrEF patients regarding clinical findings and cardiac imaging, genomics, proteomics, and transcriptomics from blood and cardiac biopsies, and by established biomarkers of fibrosis, inflammation, haemodynamics, haemostasis, and thrombosis. The data will be explored by state-of-the-art bioinformatics methods to investigate gene expression patterns, sequence variation, DNA methylation, and post-translational modifications, and using systems biology approaches including pathway and network analysis.In this epidemiological HF study with biopsy studies in a subset of patients, we aim to identify new biomarkers of disease progression and to find pathophysiological mechanisms to support explorations of new treatment regimens for HFpEF.

ELIGIBILITY:
Inclusion Criteria:CABG PREFERS

Inclusion criteria:

1. Patients undergoing elective coronary bypass surgery
2. History of heart failure not required
3. Age >18 years
4. Willingness to participate (written informed consent)
5. Possibility to obtain technically satisfactory echocardiography

Inclusion criteria PREFERS:

1. New-onset heart failure according to ESC guidelines including NT-proBNP >125 ng/L at heart failure clinic or >300 ng/L at emergency department visit or hospital admission
2. Age >18 years
3. Willingness to participate (written informed consent)
4. Possibility to obtain technically satisfactory echocardiography

Exclusion Criteria CABG PREFERS and PREFERS:

1. Cognitive impairment
2. Inability to understand Swedish language
3. Anaemia (haemoglobin level <90 g/L)
4. Heart failure primarily due to valvular disease, primary right ventricular failure, pulmonary artery hypertension, hypertrophic obstructive cardiomyopathy Infiltrative cardiomyopathy (e.g. amyloidosis, sarcoidosis, or haemochromatosis)
5. Severe co-morbidity, severe COPD, severe renal dysfunction (eGFR <30 mL/min/1.73m2). Any other co-morbid disease that will disable the ability to assess or treat heart failure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: CABG PREFERS: Patients undergoing elective coronary artery by pass surgery at the karolinska University hospital PREFERS: New onset heart failure patients at 5 hospitals in Stockholm ; Danderyds Hospital, Capio St Görans Hospital , Karolinska Solna Karolinska Huddinge, South Hospital
Sampling Method: Probability Sample
Enrollment: 683 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
Change in fibrotic biomarkers | 2 years
  For the biopsies (CABG PREFERS), the sample size is based upon the number of patients undergoing elective CABG surgery. Investigators expect to discover mRNAs from genes of potential interest in this material with relevance to differences between preserved ejection fraction, reduced ejection fraction and normal groups by bioinformatics tools. These genes will be further investigated in the blood samples of the PREFERS study and potentially in future heart biopsies. for the PREFERS new onset heart failure study. Investigators calculated a 20% difference between HFrEF and HFpEF groups with regard to both PICP and CITP (higher PICP levels and lower CITP in HFpEF vs. HFrEF) as clinically meaningful. To detect a 20% difference between the HFpEF and the HFrEF groups with 80% power and with an estimated drop-out rate of 50 patients in each group, 250 patients in each group are needed to obtain samples from 200 per group.
Reverse remodeling | 2 years
  diastolic function

SECONDARY OUTCOMES:
cardiac magnetic resonance tomography imaging | 2 years
  ECV by cMRI will be correlated to type of HF whether HFpEF or HFrEF and to echocardiographic findings

CONTACTS AND LOCATIONS:
Overall Officials: Cecilia M Linde, MD PhD, Principal Investigator — Institution of Internal medicine, Karolinska University Hospital and Karolinska Institutet
Locations (1):
- Karolinska Institutet, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Undecided
none described

REFERENCES:
- [Result] Linde C, Eriksson MJ, Hage C, Wallen H, Persson B, Corbascio M, Lundeberg J, Maret E, Ugander M, Persson H; Stockholm County/Karolinska Institutet 4D heart failure investigators. Rationale and design of the PREFERS (Preserved and Reduced Ejection Fraction Epidemiological Regional Study) Stockholm heart failure study: an epidemiological regional study in Stockholm county of 2.1 million inhabitants. Eur J Heart Fail. 2016 Oct;18(10):1287-1297. doi: 10.1002/ejhf.599. Epub 2016 Jul 7. PMID 27384611
- [Result] Asp M, Salmen F, Stahl PL, Vickovic S, Felldin U, Lofling M, Fernandez Navarro J, Maaskola J, Eriksson MJ, Persson B, Corbascio M, Persson H, Linde C, Lundeberg J. Spatial detection of fetal marker genes expressed at low level in adult human heart tissue. Sci Rep. 2017 Oct 11;7(1):12941. doi: 10.1038/s41598-017-13462-5. PMID 29021611
- [Result] Hage C, Lofgren L, Michopoulos F, Nilsson R, Davidsson P, Kumar C, Ekstrom M, Eriksson MJ, Lynga P, Persson B, Wallen H, Gan LM, Persson H, Linde C. Metabolomic Profile in HFpEF vs HFrEF Patients. J Card Fail. 2020 Dec;26(12):1050-1059. doi: 10.1016/j.cardfail.2020.07.010. Epub 2020 Aug 1. PMID 32750486
- [Derived] Lofstrom U, Linde C, Eriksson MJ, Maret E, Corbascio M, Ekstrom M, Lynga P, Wallen H, Persson B, Persson H, Hage C. Baseline characteristics and 1-year outcome by left ventricular function in the CABG PREFERS. Eur Heart J Open. 2025 Mar 5;5(2):oeaf014. doi: 10.1093/ehjopen/oeaf014. eCollection 2025 Mar. PMID 40177505
- [Derived] Cabrera C, Frisk C, Lofstrom U, Lynga P, Linde C, Hage C, Persson H, Eriksson MJ, Wallen H, Persson B, Ekstrom M. Relationship between iron deficiency and expression of genes involved in iron metabolism in human myocardium and skeletal muscle. Int J Cardiol. 2023 May 15;379:82-88. doi: 10.1016/j.ijcard.2023.03.032. Epub 2023 Mar 15. PMID 36931398
- [Derived] Linde C, Ekstrom M, Eriksson MJ, Maret E, Wallen H, Lynga P, Weden U, Cabrera C, Lofstrom U, Stenudd J, Lund LH, Persson B, Persson H, Hage C; Stockholm County/Karolinska Institutet 4D heart failure investigators. Baseline characteristics of 547 new onset heart failure patients in the PREFERS heart failure study. ESC Heart Fail. 2022 Aug;9(4):2125-2138. doi: 10.1002/ehf2.13922. Epub 2022 Apr 10. PMID 35403374